CLINICAL TRIAL: NCT01454505
Title: Safety and Efficacy of AL-53817 Nasal Spray Solution in Ragweed Sensitive Subjects in an Environmental Exposure Chamber (EEC)
Brief Title: Safety and Efficacy of AL-53817 Nasal Spray Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-10-094
Record Dates: First submitted 2011-10-17; First posted 2011-10-19 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-03

CONDITIONS: Nasal Allergies; Allergies
Keywords: Healthy subjects; Nasal allergies; Allergies; Environmental Exposure Chamber; EEC; Ragweed
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stage B/AL-53817 (Experimental): Stage B: AL-53817 nasal spray solution, 1 spray to each nostril twice a day for 4 days. On Day 5, 1 spray to each nostril 60 minutes before entering the EEC.
  Interventions: Drug: AL-53817 nasal spray solution
- Stage B/Vehicle (Placebo Comparator): Stage B: Vehicle nasal spray, 1 spray to each nostril twice a day for 4 days. On Day 5, 1 spray to each nostril 60 minutes before entering the EEC.
  Interventions: Other: Vehicle nasal spray

INTERVENTIONS:
Drug: AL-53817 nasal spray solution — Active ingredients administered in 1 of 3 concentrations during Stage A to determine maximum tolerated dose (MTD), and administered at maximum tolerated dose during Stage B.
  Arms: Stage B/AL-53817
Other: Vehicle nasal spray — Inactive ingredients used as placebo comparator during Stage A and Stage B.
  Arms: Stage B/Vehicle

SUMMARY:
The purpose of this study was to determine the maximum tolerated dose of AL-53817 (Stage A) and evaluate the safety and efficacy of AL-53817 for the treatment of allergic rhinitis (Stage B).

DETAILED DESCRIPTION:
Stage A was a 1-day, single ascending dose study utilizing 7 separate cohorts of unique subjects (healthy normal volunteers). Each cohort was administered a different dose of AL-53817 Nasal Spray Solution in order to determine the maximum tolerated dose (MTD).

In Stage B, 2 different cohorts of unique, ragweed-sensitive subjects were administered the MTD for up to 5 days twice a day to determine the safety and efficacy of AL-53817 Nasal Spray Solution for the treatment of allergic rhinitis. Subjects were required to meet minimum allergic rhinitis scores at two qualifying EEC visits to participate in the study. Subjects were continually housed in clinic during the 5-day treatment period.

ELIGIBILITY:
Stage A Inclusion Criteria:

* Willing and able to give written informed consent.
* In good health in the opinion of an appropriately qualified physician.
* Females of childbearing potential (who are not at least 1 year post-menopausal or surgically sterilized) must have a negative urine pregnancy test at Visit 1, and must not be nursing or plan to become pregnant during the course of the study.
* Other protocol-defined inclusion criteria may apply.

Stage B Inclusion Criteria:

* History of non-recalcitrant seasonal allergic rhinitis during the fall allergy season.
* Allergy to short ragweed allergen, defined by positive skin prick test for short ragweed allergen within the 12 months prior to Visit 1.
* Be in good health in the opinion of an appropriately qualified physician.
* Females of childbearing potential (who are not at least 1 year post-menopausal or surgically sterilized) must have negative urine pregnancy test at Visit 1, and must not be nursing or plan to become pregnant during the course of the study.
* Other protocol-defined inclusion criteria may apply.

Stage A Exclusion Criteria:

* Hypersensitivity to the study drug or any component of the test articles, including benzalkonium chloride.
* Using any prescription or non-prescription systemic or topical medications, vitamins or dietary supplements within 14 days prior to the check-in day (except for acetaminophen at doses of < 2 grams/day or topical, hormonal-oral, implantable or injectable contraceptives).
* Current or recent history of severe, unstable, or uncontrolled conditions based upon a review of medical history and/or physical examination.
* Any nasal disorder that could preclude safe administration of study medication and/or interfere with the evaluation of the study medication.
* History of HIV, hepatitis B or active hepatitis A as determined by medical history and/or by serology at the Screening Visit.
* Any screening clinical laboratory result (hematology, serum chemistry or urinalysis) outside the normal range that is clinically relevant in the opinion of an appropriately qualified physician and/or Alcon physician.
* Participation in any investigational study within 30 days of entry into this study or concomitantly with this study.
* Other protocol-defined exclusion criteria may apply.

Stage B Exclusion Criteria:

* Any screening clinical laboratory result (hematology, serum chemistry or urinalysis) outside the normal range that is clinically relevant in the opinion of an appropriately qualified physician and/or Alcon physician.
* Using any prescription or non-prescription systemic or topical medications, vitamins or dietary supplements within 14 days prior to the check-in day (except for acetaminophen at doses of < 2 grams/day or topical, hormonal-oral, implantable or injectable contraceptives).
* History of HIV, hepatitis B or C or active hepatitis A as determined by medical history and/or by serology at the Screening Visit.
* Any nasal disorder that could preclude safe administration of study medication and/or interfere with the evaluation of the study medication.
* Confirmed diagnosis of chronic rhinosinusitis within 12 months of Visit.
* Confirmed diagnosis of severe rhinitis or rhinosinusitis prior to Visit 1 that, in the opinion of the Investigator, would preclude safe subject participation in the study.
* Current or recent history of any severe, unstable, or uncontrolled condition that, in the opinion of the Investigator, would preclude safe participation in the study.
* Participation in any investigational study within 30 days of entry into this study or concomitantly with this study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one study center in Canada.
Pre-assignment Details: 50 healthy volunteers were enrolled in Stage A and subsequently exited from the study. 60 unique patients were enrolled in Stage B.
Groups:
- Stage A/AL-53817: AL-53817 nasal spray solution in 1 of 3 concentrations, 1 or 2 sprays per nostril, single dose
- Stage A/Vehicle: Vehicle, 1 or 2 sprays per nostril, single dose
- Stage B/AL-53817: AL-53817 nasal spray solution, 1 spray per nostril twice a day for 4 days. On Day 5, 1 spray per nostril 60 minutes before entering the EEC.
- Stage B/Vehicle: Vehicle nasal spray, 1 spray per nostril twice a day for 4 days. On Day 5, 1 spray per nostril 60 minutes before entering the EEC.
Period: Overall Study
Arm/Group | Stage A/AL-53817 | Stage A/Vehicle | Stage B/AL-53817 | Stage B/Vehicle
Started | 35 | 15 | 40 | 20
Completed | 35 | 15 | 40 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stage A/Healthy Volunteers: AL-53817 nasal spray solution in 1 of 3 concentration doses, 1 or 2 sprays per nostril, OR Vehicle, 1 spray per nostril
- Total: Total of all reporting groups
Arm/Group | Stage A/Healthy Volunteers | Stage B/AL-53817 | Stage B/Vehicle | Total
Number analyzed (Participants) | 50 | 40 | 20 | 110
Age, Customized [Number; unit: participants]
  <65 | 49 | 39 | 20 | 108
  ≥65 | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 15 | 63
  Male | 25 | 17 | 5 | 47
Region of Enrollment [Number; unit: participants]
  Canada | 50 | 40 | 20 | 110

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events in Stage A
Description: Adverse events, including serious adverse events and deaths, were reported regardless of test article relationship.
Time Frame: Day 1
Population: This reporting group includes all subjects exposed to test article during Stage A.
Measure: Number; unit: Adverse Events
Arm/Group | Stage A/AL-53817 | Stage A/Vehicle
Number analyzed (Participants) | 35 | 15
Adverse Events
  Adverse events, not including serious | 9 | 3
  Serious adverse events, not including deaths | 0 | 0
  Deaths | 0 | 0

2. Secondary Outcome: Mean Change From Baseline in Total Nasal Symptom Scores (TNSS) Over a 6-hour Period in the EEC at Day 5
Description: Stage B: Nasal symptoms were assessed by the subject before entering the EEC and at 14 timepoints over a 6-hour period after entering the EEC. TNSS score (0-12) was a sum of scores for nasal congestion, sneezing, itchy nose, and runny nose scores, each individually assessed on a 0 to 3 scale, where 0=none and 3=severe. Baseline EEC was conducted up to 21 days prior to the 5-day treatment period.
Time Frame: Baseline (pretreatment), Day 5
Population: Stage B: This reporting group includes all randomized subjects who satisfied inclusion/exclusion criteria and had EEC data at baseline and Day 5, per protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Stage B/AL-53817: AL-53817 nasal spray solution, 1 spray to each nostril twice a day for 4 days. On Day 5, 1 spray to each nostril 60 minutes before entering the EEC.
- Stage B/Vehicle: Vehicle nasal spray, 1 spray to each nostril twice a day for 4 days. On Day 5, 1 spray to each nostril 60 minutes before entering the EEC.
Arm/Group | Stage B/AL-53817 | Stage B/Vehicle
Number analyzed (Participants) | 40 | 20
Units on a scale
  0 hour | -0.3 (2.3) | 0.3 (1.7)
  0.25 hour | -0.7 (2.8) | 0.8 (2.4)
  0.5 hour | -1.5 (2.5) | 0.1 (1.8)
  0.75 hour | -2.3 (2.8) | -0.9 (2.5)
  1 hour | -2.3 (3.2) | -1.1 (2.5)
  1.5 hour | -3.1 (2.9) | -0.3 (3.5)
  2 hours | -2.8 (3.1) | -1.3 (3.2)
  2.5 hours | -2.8 (3.2) | -0.8 (3.2)
  3 hours | -2.2 (2.9) | -0.5 (2.6)
  3.5 hours | -2.9 (2.8) | -0.8 (2.9)
  4 hours | -2.7 (3.1) | -1.3 (2.6)
  4.5 hours | -2.7 (2.6) | -1.4 (3.1)
  5 hours | -2.7 (2.8) | -1.3 (2.8)
  5.5 hours | -2.7 (3.2) | -1.4 (3.4)
  6 hours | -2.3 (2.7) | -1.0 (2.8)

3. Primary Outcome: Mean Change From Baseline in Nasal Congestion Over a 6-hour Period in the EEC at Day 5
Description: Stage B: Nasal congestion was assessed by the subject before entering the EEC and at 14 timepoints over a 6-hour period after entering the EEC. Nasal congestion was scored on a scale from 0-3, where 0=none and 3=severe. Baseline EEC was conducted up to 21 days prior to the 5-day treatment period.
Time Frame: Baseline (pretreatment), Day 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Stage B/AL-53817 | Stage B/Vehicle
Number analyzed (Participants) | 40 | 20
Units on a scale
  0 hour | 0.1 (0.7) | 0.1 (0.8)
  0.25 hour | -0.1 (0.9) | 0.2 (0.8)
  0.5 hour | -0.5 (0.7) | -0.1 (0.6)
  0.75 hour | -0.6 (0.7) | -0.3 (0.7)
  1 hour | -0.6 (0.9) | -0.3 (0.6)
  1.5 hours | -0.8 (0.8) | 0.0 (1.0)
  2 hours | -0.6 (0.9) | -0.2 (1.0)
  2.5 hours | -0.7 (0.8) | -0.1 (0.8)
  3 hours | -0.5 (0.8) | -0.1 (1.0)
  3.5 hours | -0.7 (0.9) | -0.2 (0.7)
  4 hours | -0.6 (1.0) | -0.3 (1.0)
  4.5 hours | -0.7 (0.8) | -0.3 (0.9)
  5 hours | -0.7 (0.9) | -0.2 (1.0)
  5.5 hours | -0.6 (0.9) | -0.2 (1.0)
  6 hours | -0.6 (0.8) | -0.2 (0.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. This reporting group includes all subjects exposed to test article in Stage A and Stage B.
Description: An adverse event was defined as any untoward medical occurrence in a subject who was administered a study treatment regardless of whether or not the event had a causal relationship with the treatment. Adverse events were obtained as solicited comments from the subjects and as observations by the study Investigator.
Arm/Group | Stage A/AL-53817 | Stage A/Vehicle | Stage B/AL-53817 | Stage B/Vehicle
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/15 | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 5/35 | 2/15 | 31/40 | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage A/AL-53817 (N=35) | Stage A/Vehicle (N=15) | Stage B/AL-53817 (N=40) | Stage B/Vehicle (N=20)
Lacrimation increased (Eye disorders) | 1 | 0 | 3 | 0
Headache (Nervous system disorders) | 2 | 1 | 10 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 29 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 4 | 2
Respiratory rate increased (Investigations) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.